CLINICAL TRIAL: NCT03008395
Title: Empowerment, Motivation and Medical Adherence (EMMA). Dialogue Tools for Consultations With Patients With Type 2 Diabetes
Brief Title: Empowerment, Motivation and Medical Adherence (EMMA).
Acronym: EMMA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to secure clinic support for conducting research
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Michael Vallis, Lead, Behaviour Change Institute and Associate Professor, Family Medicine, Dalhousie University, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NSHABCIEMMA
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMMA (Experimental): These participants will receive diabetes self-management education using the dialogue tools, which emphasize empowerment and use the principles of motivational communication and behaviour modification. There will be a series of four visits using the dialogue tools to guide the patient toward meaningful self-management tasks. This is not the typical approach, where providers tell the patient the behaviours they, not the patient, consider priorities. This intervention will evaluate if medical outcomes (A1c) and adherence are improved using a patient-centered not a clinician-cantered approach in individuals with poor diabetes control.
  Interventions: Behavioral: EMMA
- Treatment as Usual (Active Comparator): The participants will receive standard diabetes education via group and individual sessions with certified diabetes educators. In this method the patient is provided structured education in which there is an emphasis on covering clinician-determined aspects of diabetes knowledge and self-management. The emphasis vis on diabetes educator recommendations.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: EMMA — Dialogue tools will be used to develop personally relevant behavioural goals consistent with diabetes self-management
  Arms: EMMA
Other: Treatment as Usual — Participants randomized to this intervention will receive standard diabetes education sessions. These include group education session and follow up session based on clinician-generated recommendations.
  Other Names: Standard Diabetes Education
  Arms: Treatment as Usual

SUMMARY:
Outcomes in type 2 diabetes are largely achieved by self-management efforts by individuals living with diabetes. Diabetes self-management is typically provided using the principles of adult education. Current evidence suggests that standard educational interventions are suboptimal. This study evaluates a novel approach to diabetes self-management using dialogue tools based on empowerment and motivational communication methods. The approach evaluated in this study is called EMMA: empowerment, motivation and medical adherence. Participants will be randomized to EMMA and treatment as usual, treated for a period of 4 months and evaluated over a period of 12 months.

DETAILED DESCRIPTION:
The management of type 2 diabetes (T2D) is experienced by many patients as being very complex. This is especially true when diabetes management includes multiple medical interventions such as oral agents and injectable medication (insulin, GLP-1; DPP-4s) in combination with diabetes specific behaviours such as blood glucose monitoring and foot care as well as healthy lifestyle behaviours such as physical activity and healthy eating. Studies show that 40-50 % of patients with T2D have suboptimal adherence to self-management recommendations. In general, it is estimated that about half of patients with chronic diseases do not take their medications as prescribed. Suboptimal medical adherence drives poor glycemic control as well as poor quality of life for an individual patient not to mention increased health care costs due to comorbidities, reduced work function and hospital admissions.

Suboptimal adherence may be driven by numerous factors, including lack of symptoms of TD2 (perceived nonseriousness of the disease), side-effects of treatments (GI distress associated with metformin, weight gain associated with insulin) in conjunction with a complex dosing regimen, lack of knowledge or belief in the efficiency of the medication, lack of motivation, cultural factors as well as poor instruction and judgmental communication between the healthcare professional and patient.

There is a need for new methods to understand the drivers of nonadherence and support the patient to proactively self-manage their TD2. There is also a need for new tools (i.e., knowledge translation methods) to support healthcare professionals to engage patients based on dialogue (collaboration) and active patient involvement (self-management), to overcome the barriers to adherence and thereby improve their ability to obtain good glycemic control. The purpose of this study is to evaluate a self-management support intervention called EMMA: Empowerment, motivation & medical adherence.

EMMA is a concept consisting of a number of dialogue tools for use in diabetes consultations (see below). The concept was, in its original form tested, in a feasibility study (N = 19 T2D) in 2011-12. The study showed significant reduction in HbA1c (EMMA: median decrease of 2.0 mmol / mol (-1.0 to 3.0) versus control: median increase 2.5 mmol / mol (-2.0 to -4.5) p = 0.05) (Varming 2012; Andrésdóttir 2014). The investigators have been collaborating with the Danish group who have developed the EMMA protocol and have developed training programs to support the diabetes educator in the delivery of the intervention. The use of the EMMA method is very consistent with motivational communication and behaviour change counselling. The investigators plan to conduct a small scale randomized comparison trial of the EMMA method with diabetes services at the NSHA Central Zone.

ELIGIBILITY:
Inclusion Criteria:

* Adults with type 2 diabetes ≥ 18 years
* Type 2 diabetes ≥ 1 years
* HbA1c ≥ 8 % at the last three visits before randomization
* On oral or injectable medications (insulin, GLP-1; DPP-4)
* Can speak, read and understand English

Exclusion Criteria:

* Participation in other clinical intervention studies during the trial period
* Receiving psychological or psychiatric treatment for a mental health disorder
* Severely impaired vision or blindness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 12 months
  Hemoglobin A1c is a blood test that is considered to be the gold standard of diabetes control

SECONDARY OUTCOMES:
WHO-QoL Scale | 12 months
  The validated WHO quality of life self-report index will be used to assess quality of life
Support for autonomous control over diabetes | 12 months
  The validated Healthcare Climate Questionnaire (HCCQ), measures the support for autonomy from healthcare professionals experienced by the patient
Self-management of diabetes | 12 Months
  The validated self-report scale, Treatment Self-Regulation Questionnaire (TSRQ), measures the patient's motivation for health behaviour change
Self-Efficacy at diabetes self-management | 12 Months
  The validated self-report scale, the Perceived Competence in Diabetes (PCD), measures the patient's experience of competence in diabetes self-management
Diabetes Distress | 12 Months
  The validated scale, the Diabetes Distress Scale (DDS) measures the experience of the burden of diabetes in everyday life

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vallis, PhD, Principal Investigator — Lead, Behaviour Change Institute, NSHA and Associate Professor, Family Medicine, Dalhousie University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson RM, Funnell MM, Aikens JE, Krein SL, Fitzgerald JT, Nwankwo R, Tannas CL, Tang TS. Evaluating the Efficacy of an Empowerment-Based Self-Management Consultant Intervention: Results of a Two-Year Randomized Controlled Trial. Ther Patient Educ. 2009 Jun 1;1(1):3-11. doi: 10.1051/tpe/2009002. PMID 20076768
- [Background] Aikens JE, Piette JD. Longitudinal association between medication adherence and glycaemic control in Type 2 diabetes. Diabet Med. 2013 Mar;30(3):338-44. doi: 10.1111/dme.12046. PMID 23075262
- [Background] Cushing A, Metcalfe R. Optimizing medicines management: From compliance to concordance. Ther Clin Risk Manag. 2007 Dec;3(6):1047-58. PMID 18516274
- [Background] Funnell M. Beyond the data: moving towards a new DAWN in diabetes. Diabet Med. 2013 Jul;30(7):765-6. doi: 10.1111/dme.12244. No abstract available. PMID 23710971
- [Background] Gaede P, Vedel P, Larsen N, Jensen GV, Parving HH, Pedersen O. Multifactorial intervention and cardiovascular disease in patients with type 2 diabetes. N Engl J Med. 2003 Jan 30;348(5):383-93. doi: 10.1056/NEJMoa021778. PMID 12556541
- [Background] Gaver, B, Dunne, T, Pacenti, E. Design Cultural Probes. Interactions. 1999; 6(1):21-29
- [Background] Grabowski, D, Jensen, BB, Willaing, I, Zoffmann, V, Schiøtz, M. Sundhedspædagogik in patientuddannelse. A literature-based review of selected health education principles used in patient education. 2010; Steno Diabetes Center
- [Background] Hansen, UM, Engelund, G, à Rogvi, S, Willaing, I (2014). The Balancing Person: an innovative approach to person-centered education in chronic illness. The European Journal of Person Centered Healthcare vol 2(3): 290-302
- [Background] Haynes RB, Ackloo E, Sahota N, McDonald HP, Yao X. Interventions for enhancing medication adherence. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD000011. doi: 10.1002/14651858.CD000011.pub3. PMID 18425859
- [Background] Ho PM, Rumsfeld JS, Masoudi FA, McClure DL, Plomondon ME, Steiner JF, Magid DJ. Effect of medication nonadherence on hospitalization and mortality among patients with diabetes mellitus. Arch Intern Med. 2006 Sep 25;166(17):1836-41. doi: 10.1001/archinte.166.17.1836. PMID 17000939
- [Background] Jensen ML, Jorgensen ME, Hansen EH, Aagaard L, Carstensen B. A multistate model and an algorithm for measuring long-term adherence to medication: a case of diabetes mellitus type 2. Value Health. 2014 Mar;17(2):266-74. doi: 10.1016/j.jval.2013.11.014. PMID 24636386
- [Background] Kerse N, Buetow S, Mainous AG 3rd, Young G, Coster G, Arroll B. Physician-patient relationship and medication compliance: a primary care investigation. Ann Fam Med. 2004 Sep-Oct;2(5):455-61. doi: 10.1370/afm.139. PMID 15506581
- [Background] Kvale,S. Interviews: an introduction to qualitative research interviewing. 1996. Thousand Oaks, CA; London, Sage
- [Background] Linn AJ, van Weert JC, Schouten BC, Smit EG, van Bodegraven AA, van Dijk L. Words that make pills easier to swallow: a communication typology to address practical and perceptual barriers to medication intake behavior. Patient Prefer Adherence. 2012;6:871-85. doi: 10.2147/PPA.S36195. Epub 2012 Dec 11. PMID 23271896
- [Background] Manca A, Hawkins N, Sculpher MJ. Estimating mean QALYs in trial-based cost-effectiveness analysis: the importance of controlling for baseline utility. Health Econ. 2005 May;14(5):487-96. doi: 10.1002/hec.944. PMID 15497198
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Background] Peyrot M, Rubin RR. Behavioral and psychosocial interventions in diabetes: a conceptual review. Diabetes Care. 2007 Oct;30(10):2433-40. doi: 10.2337/dc07-1222. Epub 2007 Jul 31. No abstract available. PMID 17666457
- [Background] Rhee MK, Slocum Pawson & Tilley. Realistic Evaluation. 1997. London: Sage
- [Background] Rhee MK, Slocum W, Ziemer DC, Culler SD, Cook CB, El-Kebbi IM, Gallina DL, Barnes C, Phillips LS. Patient adherence improves glycemic control. Diabetes Educ. 2005 Mar-Apr;31(2):240-50. doi: 10.1177/0145721705274927. PMID 15797853
- [Background] Richard C, Lussier MT. MEDICODE: an instrument to describe and evaluate exchanges on medications that occur during medical encounters. Patient Educ Couns. 2006 Dec;64(1-3):197-206. doi: 10.1016/j.pec.2006.02.002. Epub 2006 Jun 16. PMID 16782298
- [Background] Skinner TC, Carey ME, Cradock S, Dallosso HM, Daly H, Davies MJ, Doherty Y, Heller S, Khunti K, Oliver L; DESMOND Collaborative. 'Educator talk' and patient change: some insights from the DESMOND (Diabetes Education and Self Management for Ongoing and Newly Diagnosed) randomized controlled trial. Diabet Med. 2008 Sep;25(9):1117-20. doi: 10.1111/j.1464-5491.2008.02492.x. PMID 19183318
- [Background] Tang TS, Funnell MM, Gillard M, Nwankwo R, Heisler M. The development of a pilot training program for peer leaders in diabetes: process and content. Diabetes Educ. 2011 Jan-Feb;37(1):67-77. doi: 10.1177/0145721710387308. Epub 2011 Jan 10. PMID 21220362
- [Background] Teasdale, T & Svendsen, H. Psykologiske & pædagogiske metoder. Kvalitative og kvantitative forskningsmetoder I praksis. Jensen T.B. and Christensen G (eds.). 2005. Frederiksberg:Roskilde Universitetsforla
- [Background] van Dulmen S. The value of tailored communication for person-centred outcomes. J Eval Clin Pract. 2011 Apr;17(2):381-3. doi: 10.1111/j.1365-2753.2010.01586.x. Epub 2010 Nov 18. PMID 21087372
- [Background] Vallis M. Behaviour change counselling--how do I know if I am doing it well? The development of the Behaviour Change Counselling Scale (BCCS). Can J Diabetes. 2013 Feb;37(1):18-26. doi: 10.1016/j.jcjd.2013.01.005. Epub 2013 Mar 14. PMID 24070744
- [Background] Varming, A. Development and usability of a participatory adherence programme aimed at patients with type 2 diabetes in poor glycemic control. 2012. Master thesis (Master of Drug Management), University of Copenhagen
- [Background] Varming, A., Andrésdóttir, G., Engelund, G., Jelstrup, L., Persson, F. I. EMMA: Empowerment, Motivation & Medical Adherence. Dialogue tools for diabetes consultations. ISBN 978-87-92759-07-8. Steno Diabetes Center. 2013 Gentofte.
- [Background] Williams A, Manias E, Walker R. Interventions to improve medication adherence in people with multiple chronic conditions: a systematic review. J Adv Nurs. 2008 Jul;63(2):132-43. doi: 10.1111/j.1365-2648.2008.04656.x. PMID 18537843
- [Background] World Health Organization. Adherence to long-term therapies: evidence for action. 2003